CLINICAL TRIAL: NCT03361111
Title: Utility of Biomarkers in Evaluating Responsiveness to Anti-IgE (Omalizumab) in Severe Asthma Patients
Brief Title: BIOmarkers in Severe AsthMa Patients on Omalizumab Treatment
Acronym: BIOSAMOT
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Joanna Hermanowicz-Salamon, MD PhD, Medical University of Warsaw
Other Study IDs: Dep. of Pneum. and Allerg.
Record Dates: First submitted 2017-11-12; First posted 2017-12-04 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Severe Asthma
Keywords: severe asthma; anti-IgE; periostin; induced sputum,; exhaled breath condensate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophil infiltration and degranulation in airways has been implicated in the pathology of asthma. Periostin is considered to be a marker of eosinophilic inflammation and is one of the highly expressed genes in epithelial cells and lung fibroblasts in asthma. Omalizumab is approved as add-on therapy in the treatment of severe allergic asthma. The aim of the study is to assess inflammatory biomarkers including: blood and sputum eosinophilia, periostin and IL-6 as long-term clinical outcomes of omalizumab therapy.

DETAILED DESCRIPTION:
Anti-IgE (omalizumab) has been shown to be an effective add-on therapy for patients with allergic severe asthma. In this observational study patients aged over 18 year with uncontrolled severe persistent asthma are selected for add-on therapy with omalizumab. Patients were on high dose of ICS and had a documented history of 2-6 exacerbations requiring treatment with systemic corticosteroids ( with >15 mg/day prednisone or other medications at similar dose, for at least 3 days). The individual dose and frequency of omalizumab administration is assessed from the dosing table. Lung function tests and asthma questionnaires (ACQ, AQLQ and RQLQ) are used in the aim of assessing clinical improvement after omalizumab treatment. Induced sputum (IS) and exhaled breath condensate (EBC) are used as a simple non-invasive methods for monitoring cellular and biochemical changes in the airways. Total blood eosinophil count, IS cytology, IS and EBC periostin and IL-6 concentrations are measured. Analyses are performed at entry and after 16, 52 and 104,156 weeks of omalizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. positive history of atopy
2. serum total IgE level between 30 and 700 IU/ml
3. body weight not more than 150 kg
4. high dose of ICS and LABA
5. a documented history of 2-6 exacerbations requiring treatment with systemic corticosteroids ( with >15 mg/day prednisone or other medications at similar dose, for at least 3 days).

Exclusion Criteria:

1. smoking
2. pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe allergic asthma
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in selected biomarkers in induced sputum | baseline and after 156 weeks of omalizumab treament
  eosinophil count
Change in selected biomarkers in peripheral blood | baseline and after 156 weeks of omalizumab treament
  eosinophil count
Change in selected biomarkers in induced sputum | baseline and after 156 weeks of omalizumab treament
  periostin
Change in selected biomarkers in exhaled breath condensate | baseline and after 156 weeks of omalizumab treament
  periostin
Change in selected biomarkers in induced sputum | baseline and after 156 weeks of omalizumab treament
  IL-6
Change in selected biomarkers in exhaled breath condensate | baseline and after 156 weeks of omalizumab treament
  IL-6

SECONDARY OUTCOMES:
Change in selected biomarkers in induced sputum | baseline and after at 16,52,104 weeks of omalizumab treament
  eosinophils, periostin, IL-6
Change in selected biomarkers in exhaled breath condensate | baseline and after at 16, 52, 104 weeks of omalizumab treament
  periostin, IL-6
Change in selected biomarkers in peripheral blood | baseline and after at 16, 52, 104 weeks of omalizumab treament
  eosinophil count

OTHER OUTCOMES:
Lung function tests | baseline and after at 16, 52, 104, 156 weeks of treament
  FEV1, FVC, FEV1/FVC

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Hermanowicz-Salamon, MD,PhD, Principal Investigator — Department of Internal Medicine, Pulmonary Diseases and Allergy Medical University of Warsaw, Poland
Locations (1):
- Joanna Hermanowicz-Salamon, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodrigo GJ, Neffen H, Castro-Rodriguez JA. Efficacy and safety of subcutaneous omalizumab vs placebo as add-on therapy to corticosteroids for children and adults with asthma: a systematic review. Chest. 2011 Jan;139(1):28-35. doi: 10.1378/chest.10-1194. Epub 2010 Aug 5. PMID 20688929
- [Result] Hanania NA, Wenzel S, Rosen K, Hsieh HJ, Mosesova S, Choy DF, Lal P, Arron JR, Harris JM, Busse W. Exploring the effects of omalizumab in allergic asthma: an analysis of biomarkers in the EXTRA study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):804-11. doi: 10.1164/rccm.201208-1414OC. PMID 23471469
- [Result] ten Brinke A, Zwinderman AH, Sterk PJ, Rabe KF, Bel EH. Factors associated with persistent airflow limitation in severe asthma. Am J Respir Crit Care Med. 2001 Sep 1;164(5):744-8. doi: 10.1164/ajrccm.164.5.2011026. PMID 11549526
- [Result] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Result] Jia G, Erickson RW, Choy DF, Mosesova S, Wu LC, Solberg OD, Shikotra A, Carter R, Audusseau S, Hamid Q, Bradding P, Fahy JV, Woodruff PG, Harris JM, Arron JR; Bronchoscopic Exploratory Research Study of Biomarkers in Corticosteroid-refractory Asthma (BOBCAT) Study Group. Periostin is a systemic biomarker of eosinophilic airway inflammation in asthmatic patients. J Allergy Clin Immunol. 2012 Sep;130(3):647-654.e10. doi: 10.1016/j.jaci.2012.06.025. Epub 2012 Aug 1. PMID 22857879